CLINICAL TRIAL: NCT01009580
Title: A 26-week, Randomised, Open-labelled, Two-arm, Parallel-group, Treat-to-target Trial Comparing Efficacy and Safety of Soluble Insulin Analogue Combination (SIAC) Twice Daily (BID) With Biphasic Insulin Aspart (BIAsp) 30 BID, With or Without Metformin, With or Without DPP-4 Inhibitor, With or Without Pioglitazone in Subjects With Type 2 Diabetes in Inadequate Glycaemic Control on Once or Twice Daily Premixed or Self-mixed Insulin Regimen With or Without OADs (BOOST™: Intensify Premix 1)
Brief Title: Comparison of NN5401 With Biphasic Insulin Aspart 30 in Type 2 Diabetes
Acronym: BOOST™
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN5401-3592; 2008-005768-15 (EudraCT Number); U1111-1111-8545 (Other: WHO)
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Results first posted 2015-11-20 (Estimated); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — insulin degludec, insulin aspart drug combination; insulin aspart, insulin aspart protamine drug combination 30:70

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- IDegAsp BID (Experimental)
  Interventions: Drug: insulin degludec/insulin aspart
- BIAsp 30 BID (Experimental)
  Interventions: Drug: biphasic insulin aspart 30

INTERVENTIONS:
Drug: insulin degludec/insulin aspart — Injected s.c. (under the skin) with the breakfast meal and main evening meal. The dose were individually adjusted. Subjects continued their pre-trial OADs (oral antidiabetic drug(s)) treatment of Metformin, the specific DPP-4 Inhibitor and Pioglitazone.
  Arms: IDegAsp BID
Drug: biphasic insulin aspart 30 — Injected s.c. (under the skin) with the breakfast meal and main evening meal. The dose were individually adjusted. Subjects continued their pre-trial OADs (oral antidiabetic drug(s)) treatment of Metformin, the specific DPP-4 Inhibitor and Pioglitazone.
  Arms: BIAsp 30 BID

SUMMARY:
This trial is conducted in Asia, Europe and Oceania. The aim of this clinical trial is to compare NN5401 (insulin degludec/insulin aspart) with biphasic insulin aspart 30 in subjects with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus (diagnosed clinically) for at least 6 months
* Subjects on premixed human or analogue insulin or self-mixed insulin regimen, containing 20-40 % fast/rapid-acting component, once daily (OD) or twice daily (BID), with or without oral antidiabetic drugs) (OADs) (metformin, sulphonylurea (SU), glinides, alpha-glucosidase inhibitor, DPP-4 (dipeptidyl peptidase-4) inhibitor and pioglitazone), for at least 3 months before Visit 1
* HbA1c 7.0-10.0 % (both inclusive) by central laboratory analysis
* Body Mass Index (BMI) below or equal to 40.0 kg/m^2

Exclusion Criteria:

* Treatment with other insulin regimens than those listed in key inclusion criterion no. 2 within 3 months
* Treatment with rosiglitazone or glucagon-like peptide-1 (GLP-1) receptor agonists (exenatide, liraglutide) within 3 months prior to visit 1
* Cardiovascular disease within the last 6 months prior to visit 1, defined as: stroke; decompensated heart failure New York Heart Association (NYHA) class III or IV; myocardial infarction; unstable angina pectoris; or coronary arterial bypass graft or angioplasty
* Uncontrolled treated/untreated severe hypertension (systolic blood pressure at least 180 millimetre (mm) mercury (Hg) and/or diastolic blood pressure at least 100 mmHg)
* Pregnancy, breast-feeding, the intention of becoming pregnant or not using adequate contraceptive measures according to local requirements
* Cancer and medical history of cancer (except basal cell skin cancer and squamous cell skin cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 447 (Actual)
Dates: Start 2009-11-05 (Actual); Primary Completion 2010-08-23 (Actual); Study Completion 2010-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (47):
- Australia (5):
  - Novo Nordisk Investigational Site, St Leonards, New South Wales
  - Novo Nordisk Investigational Site, Wollongong, New South Wales
  - Novo Nordisk Investigational Site, East Ringwood, Victoria
  - Novo Nordisk Investigational Site, Melbourne, Victoria
  - Novo Nordisk Investigational Site, Garran
- Denmark (7):
  - Novo Nordisk Investigational Site, Århus C
  - Novo Nordisk Investigational Site, Copenhagen
  - Novo Nordisk Investigational Site, Gentofte Municipality
  - Novo Nordisk Investigational Site, Hjørring
  - Novo Nordisk Investigational Site, Horsens
  - Novo Nordisk Investigational Site, Hvidovre
  - Novo Nordisk Investigational Site, Svendborg
- Finland (5):
  - Novo Nordisk Investigational Site, Kuopio
  - Novo Nordisk Investigational Site, Lahti
  - Novo Nordisk Investigational Site, Oulu
  - Novo Nordisk Investigational Site, Pori
  - Novo Nordisk Investigational Site, Ylitornio
- India (8):
  - Novo Nordisk Investigational Site, Karnāl, Haryana
  - Novo Nordisk Investigational Site, Bangalore, Karnataka
  - Novo Nordisk Investigational Site, Trivandrum, Kerala
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, Chennai, Tamil Nadu
  - Novo Nordisk Investigational Site, Kolkata
  - Novo Nordisk Investigational Site, Mumbai
  - Novo Nordisk Investigational Site, New Delhi
- Malaysia (4):
  - Novo Nordisk Investigational Site, Cheras
  - Novo Nordisk Investigational Site, Kota Bharu, Kelantan
  - Novo Nordisk Investigational Site, Pulau Pinang
  - Novo Nordisk Investigational Site, Putrajaya
- Poland (6):
  - Novo Nordisk Investigational Site, Bialystok
  - Novo Nordisk Investigational Site, Bydgoszcz
  - Novo Nordisk Investigational Site, Gniewkowo
  - Novo Nordisk Investigational Site, Płock
  - Novo Nordisk Investigational Site, Rawa Mazowiecka
  - Novo Nordisk Investigational Site, Warsaw
- Sweden (5):
  - Novo Nordisk Investigational Site, Falun
  - Novo Nordisk Investigational Site, Karlstad
  - Novo Nordisk Investigational Site, Lund
  - Novo Nordisk Investigational Site, Malmo
  - Novo Nordisk Investigational Site, Stockholm
- Taiwan (3):
  - Novo Nordisk Investigational Site, Changhua
  - Novo Nordisk Investigational Site, Chiayi City
  - Novo Nordisk Investigational Site, Taipei
- Thailand (2):
  - Novo Nordisk Investigational Site, Bangkok
  - Novo Nordisk Investigational Site, Chiang Mai
- Turkey (Türkiye) (2):
  - Novo Nordisk Investigational Site, Istanbul
  - Novo Nordisk Investigational Site, Kocaeli

REFERENCES:
- [Background] Evans M, Gundgaard J, Hansen BB. Cost-Effectiveness of Insulin Degludec/Insulin Aspart Versus Biphasic Insulin Aspart in Patients with Type 2 Diabetes from a Danish Health-Care Perspective. Diabetes Ther. 2016 Dec;7(4):809-823. doi: 10.1007/s13300-016-0195-6. Epub 2016 Aug 23. PMID 27553066
- [Result] Fulcher GR, Christiansen JS, Bantwal G, Polaszewska-Muszynska M, Mersebach H, Andersen TH, Niskanen LK; BOOST: Intensify Premix I Investigators. Comparison of insulin degludec/insulin aspart and biphasic insulin aspart 30 in uncontrolled, insulin-treated type 2 diabetes: a phase 3a, randomized, treat-to-target trial. Diabetes Care. 2014 Aug;37(8):2084-90. doi: 10.2337/dc13-2908. Epub 2014 May 8. PMID 24812432
- [Result] Christiansen JS, Niskanen L, Rasmussen S, Johansen T, Fulcher G. Lower rates of hypoglycemia during maintenance treatment with insulin degludec/insulin aspart versus biphasic insulin aspart 30: a combined analysis of two Phase 3a studies in type 2 diabetes. J Diabetes. 2016 Sep;8(5):720-8. doi: 10.1111/1753-0407.12355. Epub 2016 Mar 6. PMID 26612062
- [Result] Haluzik M, Fulcher G, Pieber TR, Bardtrum L, Tutkunkardas D, Rodbard HW. The co-formulation of insulin degludec and insulin aspart lowers fasting plasma glucose and rates of confirmed and nocturnal hypoglycaemia, independent of baseline glycated haemoglobin levels, disease duration or body mass index: A pooled meta-analysis of phase III studies in patients with type 2 diabetes. Diabetes Obes Metab. 2018 Jul;20(7):1585-1592. doi: 10.1111/dom.13261. Epub 2018 Mar 25. PMID 29451706
- [Result] Fulcher G, Mehta R, Fita EG, Ekelund M, Bain SC. Efficacy and Safety of IDegAsp Versus BIAsp 30, Both Twice Daily, in Elderly Patients with Type 2 Diabetes: Post Hoc Analysis of Two Phase 3 Randomized Controlled BOOST Trials. Diabetes Ther. 2019 Feb;10(1):107-118. doi: 10.1007/s13300-018-0531-0. Epub 2018 Nov 24. PMID 30474818
- [Derived] Yang W, Akhtar S, Franek E, Haluzik M, Hirose T, Kalyanam B, Kar S, Wu T, Gogas Yavuz D, Unnikrishnan AG. Postprandial Glucose Excursions in Asian Versus Non-Asian Patients with Type 2 Diabetes: A Post Hoc Analysis of Baseline Data from Phase 3 Randomised Controlled Trials of IDegAsp. Diabetes Ther. 2022 Feb;13(2):311-323. doi: 10.1007/s13300-021-01196-7. Epub 2022 Jan 19. PMID 35044568
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial was conducted at 50 sites in 10 countries: Australia (5 sites), Denmark (7 sites), Finland (5 sites), India (9 sites), Malaysia (3 sites), Poland (5 sites), Sweden (6 sites), Taiwan (3 sites), Thailand (3 sites), Turkey (4 sites).
  In addition, 1 site in Thailand screened but did not randomise any subjects.
Pre-assignment Details: Between screening and randomisation, eligible subjects were to continue their usual pre-trial oral anti-diabetic drug (OAD) of metformin, pioglitazone and DPP-4 inhibitor.
Groups:
- IDegAsp BID: Insulin degludec/insulin aspart (IDegAsp) was given subcutaneously twice daily (BID) with or without Metformin, DPP-4 inhibitor, Pioglitazone. IDegAsp was given with the breakfast meal and main evening meal.
- BIAsp 30 BID: Biphasic insulin aspart 30 (BIAsp 30) was given subcutaneously twice daily (BID) with or without Metformin, DPP-4 inhibitor, Pioglitazone. BIAsp 30 was given with the breakfast meal and main evening meal.
Period: Overall Study
Arm/Group | IDegAsp BID | BIAsp 30 BID
Started | 224 | 223
Exposed | 224 | 222 (One subject was randomised in error and withdrew prior to exposure to drug)
Completed | 197 | 188
Not Completed | 27 | 35
Not completed — Adverse Event | 4 | 4
Not completed — Lack of Efficacy | 0 | 1
Not completed — Protocol Violation | 2 | 3
Not completed — Withdrawal Criteria | 4 | 6
Not completed — Unclassified | 17 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | IDegAsp BID | BIAsp 30 BID | Total
Number analyzed (Participants) | 224 | 222 | 446
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.7 (9.9) | 58.8 (9.8) | 58.7 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 103 | 198
  Male | 129 | 119 | 248
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.3 (0.8) | 8.4 (0.9) | 8.4 (0.8)
Fasting plasma glucose (FPG) [Mean (Standard Deviation); unit: mmol/L] | 8.9 (2.9) | 8.6 (2.6) | 8.7 (2.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycosylated Haemoglobin (HbA1c)
Description: Change from baseline in HbA1c after 26 weeks of treatment.
Time Frame: Week 0, Week 26
Population: The full analysis set (FAS) included all randomised subjects and missing data were imputed using last observation carried forward (LOCF). One subject was randomised in error, hence removed from the FAS.
Measure: Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 224 | 222
percentage of glycosylated haemoglobin | -1.28 (0.94) | -1.30 (0.97)

2. Secondary Outcome: Mean of 9-point Self Measured Plasma Glucose Profile (SMPG)
Description: Mean of SMPG after 26 weeks of treatment. Plasma glucose measured: before breakfast, 90 minutes after start of breakfast, before lunch, 90 minutes after start of lunch, before dinner, 90 minutes after start of dinner, bedtime, at 4 am and before breakfast.
Time Frame: Week 26
Population: The full analysis set (FAS) included all randomised subjects and missing data were imputed using last observation carried forward (LOCF). One subject was randomised in error, hence removed from the FAS. For 24 subjects all 9-point SMPG values were missing.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 211 | 211
mmol/L | 7.0 (1.6) | 7.3 (2.1)

3. Secondary Outcome: Rate of Confirmed Hypoglycaemic Episodes
Description: Rate of confirmed hypoglycaemic episodes per 100 patient years of exposure (PYE). Confirmed hypoglycaemic episodes consisted of severe hypoglycaemia as well as minor hypoglycaemic episodes. Severe hypoglycaemic episodes were defined as requiring assistance to administer carbohydrate, glucagon, or other resuscitative actions. Minor hypoglycaemic episodes were defined as able to treat her/himself and plasma glucose below 3.1 mmol/L.
Time Frame: Week 0 to Week 26 + 7 days follow up
Population: The safety analysis set included all subjects who received at least one dose of the investigational product or its comparator.
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 224 | 222
Episodes/100 years of patient exposure | 972 | 1396

4. Secondary Outcome: Rate of Nocturnal Confirmed Hypoglycaemic Episodes
Description: Rate of confirmed hypoglycaemic episodes per 100 patient years of exposure (PYE). Confirmed hypoglycaemic episodes consisted of severe hypoglycaemia as well as minor hypoglycaemic episodes. Severe hypoglycaemic episodes were defined as requiring assistance to administer carbohydrate, glucagon, or other resuscitative actions. Minor hypoglycaemic episodes were defined as able to treat her/himself and plasma glucose below 3.1 mmol/L. Nocturnal hypoglycaemic episodes were defined as occurring between 00:01 and 05:59 a.m.
Time Frame: Week 0 to Week 26 + 7 days follow up
Population: as for outcome 3
Measure: Number; unit: Episodes/100 years of patient exposure
Arm/Group | IDegAsp BID | BIAsp 30 BID
Number analyzed (Participants) | 224 | 222
Episodes/100 years of patient exposure | 74 | 253

ADVERSE EVENTS:
Time Frame: The adverse events were collected in a time frame of 26 weeks + 7 days follow up
Description: The safety analysis set included all subjects who received at least one dose of the investigational product or its comparator.
Arm/Group | IDegAsp BID | BIAsp 30 BID
Serious Adverse Events (participants affected / at risk) | 19/224 | 36/222
Other Adverse Events (participants affected / at risk) | 60/224 | 52/222
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDegAsp BID (N=224) | BIAsp 30 BID (N=222)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Angina unstable (Cardiac disorders) | 0 (0) | 1 (1)
Arrhythmia supraventricular (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac asthma (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0)
Diabetic retinopathy (Eye disorders) | 0 (0) | 2 (2)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2)
Malaria (Infections and infestations) | 0 (0) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Vestibular neuronitis (Infections and infestations) | 1 (1) | 1 (1)
Alcohol poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incorrect dose administered (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radius fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Snake bite (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (3) | 6 (6)
Hypoglycaemic unconsciousness (Metabolism and nutrition disorders) | 0 (0) | 5 (5)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carpal tunnel syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cervicobrachial syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Adenomyosis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Intermittent claudication (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDegAsp BID (N=224) | BIAsp 30 BID (N=222)
Pyrexia (General disorders) | 13 (15) | 0 (0)
Nasopharyngitis (Infections and infestations) | 26 (28) | 21 (28)
Upper respiratory tract infection (Infections and infestations) | 17 (19) | 17 (18)
Headache (Nervous system disorders) | 13 (16) | 18 (22)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Novo Nordisk maintains the right to be informed of any Investigator plans for publication and to review any scientific paper, presentation, communication or other information concerning the investigation described in this protocol. Any such communication must be submitted in writing to the Novo Nordisk trial manager prior to submission for comments. Comments will be given within four weeks from receipt of the planned communication.